CLINICAL TRIAL: NCT07198204
Title: Effect of Isometric Exercise Duration on Muscle Strength, Pain, and Function in Patients With Knee Osteoarthritis: A Randomized Controlled Trial
Brief Title: Different Hold Durations in Isometric Exercises
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hail (Other)
Responsible Party: Principal Investigator, Hisham Mohamed Hussein, Associate Professor, University of Hail
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FPTBSUREC/1207/14925
Record Dates: First submitted 2025-09-15; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Knee Arthritis Osteoarthritis
Keywords: knee; arthritis; strength; contraction time; isometric
MeSH Terms: conditions — Arthritis | interventions — Exercise; Ultrasonic Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- group 1 (Experimental): The subjects in this group will perform isometric exercises, including isometric quadriceps, straight-leg raising, and isometric hip adduction exercises for 5 seconds.
  All exercises will be performed in sets of 12 repetitions: one set twice a day for the 1st week, which will be progressed weekly until three sets twice a day by 3th week. Allow 5 seconds of rest between each repetition and 3 minutes of rest between sets, with a total contraction time of 60 to 180 seconds per session at 30 to 50% of maximum voluntary contraction (MVC).
  Interventions: Other: isometric exercises; Other: therapeutic ultrasound; Other: Transcutanous electrical nerve stimulation
- group 2 (Experimental): The subjects in this group will perform isometric exercises, including isometric quadriceps, straight leg raising, and isometric hip adduction exercise for 10 sec.
  All exercises will be performed in sets of 6 repetitions: one set twice a day for the 1st week, which will be progressed weekly until three sets twice a day by 3th week. Allow 10 seconds of rest between each repetition and 3 minutes of rest between sets, with a total contraction time of 60 to 180 seconds per session at 30 to 50% of MVC.
  Interventions: Other: isometric exercises; Other: therapeutic ultrasound; Other: Transcutanous electrical nerve stimulation
- group 3 (Experimental): The subjects in this group will perform isometric exercises, including isometric quadriceps, straight leg raising, and isometric hip adduction exercise for 20 sec.
  All exercises will be performed in sets of 3 repetitions: one set twice a day for the 1st week, which will be progressed weekly until three sets twice a day by 3th week. Allow 20 seconds of rest between each repetition and 3 minutes of rest between sets, with a total contraction time of 60 to 180 seconds per session at 30 to 50% of MVC.
  Interventions: Other: isometric exercises; Other: therapeutic ultrasound; Other: Transcutanous electrical nerve stimulation
- control group (Active Comparator): The control group will receive ultrasound therapy and TENS only.
  Interventions: Other: therapeutic ultrasound; Other: Transcutanous electrical nerve stimulation

INTERVENTIONS:
Other: isometric exercises — Isometric quadriceps exercise: Patients lie in a supine position. A rolled-up towel was put beneath the knee. They were instructed to maximally activate their thigh muscles to straighten their knee and hold the contraction for 5 seconds (Group A), 10 seconds (Group B), or 20 seconds (Group C).
  Arms: group 1; group 2; group 3
Other: therapeutic ultrasound — all patients will reciece ultrasound for 5 minutes using 1MHz frequency, 0.8 wc2, 5cm2 head with adequate gel as a coupling medium
Other: Transcutanous electrical nerve stimulation — all participants will recieve TENS for 30 minutes per session. the parameters will be Burst TENS, with main frequency of 100Hz, burst frequency of 4 Hz, intensity to the comfortable muscle twitch, electrodes size according to the size of the patients knee.

SUMMARY:
this stuy tries to evaulate the best contraction (hold time) during isometric effort that can provide the best therapeutic effects on muscular performance in patients with knee osteoarthritis

DETAILED DESCRIPTION:
Knee osteoarthritis (KOA) is a common degenerative disease characterized by the gradual degeneration and loss of joint cartilage, accompanied by bone proliferation. These pathological changes lead to joint pain, stiffness, and limited mobility in affected individuals (Sharma, 2021). The development of KOA, usually associated with various risk factors including age, gender, obesity, genetics, and joint injuries, severely affects patients' quality of life and imposes a heavy economic burden on society (Katz et al., 2021). Research indicates that the global prevalence of KOA has increased significantly since 1990 and is expected to continue rising until 2050, posing a major challenge to global public health.(Steinmetz et al., 2023) Currently, there are various treatment methods for KOA, including pharmacotherapy, surgical treatment, and physical therapy (Duong et al., 2023). Although pharmacotherapy can effectively alleviate symptoms, long-term use may lead to a series of side effects.

Due to its low impact and reduced joint stress, isometric exercise may be more suitable for patients sensitive to joint stress or at higher risk; however, the optimal duration for isometric exercises remains controversial and varies. For instance, Folland et al. compared the strength gains produced by isometric training (with contraction duration of 2 seconds) at four joint angles with conventional dynamic training(Folland et al., 2005). In another study, Kubo et al. investigated the effects of static and dynamic training on the stiffness and blood volume of the human tendon, using a training regimen of 10 contractions of 15-s duration for isometric knee extensions (Kubo et al., 2009). Additionally, Anwer & Alghadir utilized a 5-second duration for isometric quadriceps contractions and hip adduction exercises. In contrast, the Straight Leg Raising (SLR) exercise was maintained for a contraction time of 10 seconds to assess the effects of isometric quadriceps exercises on individuals with knee osteoarthritis.

Understanding the isometric exercise parameters, such as duration, that achieve a desired adaptive response in muscle and tendon would benefit optimizing results. Therefore, the purpose of this study is to compare the effect of isometric exercise duration on muscle strength, pain, and function in patients with KOA.

ELIGIBILITY:
Inclusion Criteria:

* prediagnosed case of knee OA as per the American College of Rheumatology (ACR) and radiological evidence of primary osteoarthritis of grade 3 or less on the Kellgren Lawrence scale;
* age between 40-65 years, including both men and women.
* unilateral or bilateral involvement (in the case of bilateral involvement, the more symptomatic knee was included).

Exclusion Criteria:

* Other knee joint pathologies, eg, Chondromalacia patella, plica syndrome,
* Neurological disorders.
* Patients having lower extremity injury/surgeries in the past 6 months,
* Hip or knee fractures or deformity,
* joint infections and inflammatory joint disease,
* physical therapy on the knee within the last 3 months or steroid injections,

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-11-30 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
pain by numeric pain rating scale | at baseline and after 1month of trreatment
  The Numeric Pain Rating Scale (NPRS) is the simplest and most commonly used numeric scale to rate pain, ranging from 0 (no pain) to 10 (worst pain). The NPRS will be used for subjective pain measurement, which has good test-retest reliability
Function using Western Ontario and McMaster Universities Osteoarthritis | will be assessed at baseline and after 1 month of treatement
  We will focus only on stiffness and physical function. The Western Ontario and McMaster Universities Osteoarthritis (WOMAC) has been widely used by clinicians in assessing patients with knee OA since it was developed in 1986 (Bellamy, 1995) to evaluate the symptoms of pain, stiffness, and physical function in patients with hip and/or knee OA. It consists of 24 questions and is divided into 3 subgroups: the pain subgroup consists of 5 questions, the stiffness subgroup consists of 2 questions, and the physical function subgroup consists of 17 questions. Each question receives a value between 0 and 4, and the total score is calculated as follows: no difficulty is scored as 0, mild as 1, moderate as 2, severe as 3, and extreme as 4. Higher scores indicate greater physical dysfunction and disability, and thereby worse health-related quality of life
function using Five Times Sit to Stand Test | at baseline and after 1month of treatment
  The muscle strength of the lower limbs was measured by the Five-Times-Sit-to-Stand Test (FTSST), in which participants rise from a chair and return to a seated position as quickly as possible with their arms folded across their chests. The time to complete five repetitions was recorded for two separate trials, with a 1-minute rest between each trial. The mean of the two trials was computed and used in the analysis
muscle strength using the one-repetition maximum (1RM) test for knee extension | at baseline and after 1 month of treatement
  1RM test has good-to-excellent test-retest reliability. the participants will be asked to perform active knee extension against different pregressive increasing weigths to determine the 1 RM. 2 minutes rest will be allowed before each contraction effort to allow recovery of the tested muscle.

IPD SHARING:
Plan to Share IPD: No
data will be used in future research